CLINICAL TRIAL: NCT04052971
Title: A Phase 1 Multicenter, Open-Label, Dose-Escalation Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of ABN401 in Patients With Advanced Solid Tumors and Pilot Expansion in Patients With Non-Small Cell Lung Cancer Harboring c-MET Dysregulation
Brief Title: To Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of ABN401 in Patients With Advanced Solid Tumors and Non-Small Cell Lung Cancer Harboring c-MET Dysregulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abion Inc (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABN401-001
Record Dates: First submitted 2019-07-26; First posted 2019-08-12 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Escalation phase (Experimental): Drug: ABN401
  Route of Administration: Oral
  The study will follow a single patient cohort approach for the first 3 regular dose levels followed by classic 3+3 design. The starting dose is 50mg QD.
  Interventions: Drug: ABN401- Escalation Phase
- Expansion phase (Experimental): Drug: ABN401
  Route of Administration: Oral
  Once the maximum tolerated dose (MTD) or highest escalation cohort has been reached, or notable efficacy has been observed at a given dose level, a decision as to Recommended Phase 2 dose (RP2D) will be determined. Up to 40 patients with Non-Small Cell Lung Cancer Harboring c-MET Dysregulation will be recruited.
  Interventions: Drug: ABN401- Expansion Phase

INTERVENTIONS:
Drug: ABN401- Escalation Phase — Dose administration: Escalation Phase The regular dose levels of ABN401 will range from 50 mg to 1800 mg QD daily for 21 days.
  Arms: Escalation phase
Drug: ABN401- Expansion Phase — Dose administration: Expansion Phase The expansion phase of the study will use the dose and schedule determined to be most appropriate in the dose escalation portion of the study. This may be the MTD and/or the RP2D and will consist of cohorts of NSCLC patients with c-MET dysregulation.
  Patients will receive ABN401 800 mg, administered orally once daily for 21 days until disease progression, unacceptable toxicity, or patient withdrawal.
  Arms: Expansion phase

SUMMARY:
This is a dose escalation, Phase 1 study of ABN401 in patients with advanced solid tumors, refractory metastatic disease, or refractory locally advanced disease not amenable to local therapy.

DETAILED DESCRIPTION:
First part of the study uses single patient cohorts at the initial dose levels, followed by a classic 3+3 design, with enrollment of 3 patients per cohort and expansion to 6 patients in the event of a dose-limiting toxicity (DLT).

The second part of the study consists of expansion cohorts will enroll Non-Small Cell Lung Cancer Harboring patients with c-MET dysregulation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent before any study-specific screening procedures.
2. Male or female ≥ 18 years of age or designated age of majority according to regulatory authorities, whichever is higher.
3. Body weight ≥ 40 kg and ≤ 110 kg.
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS), 0 or 1.
5. Diagnosis:

   1. For the Phase 1 dose escalation, must have:

      * Histological or cytological diagnosis of melanoma or any type of carcinoma or sarcoma,
      * Refractory metastatic disease, or refractory locally advanced disease not amenable to local therapy,
      * Metastatic breast or prostate cancer may have bone-only disease.
   2. For the Phase 1 extension (pilot expansion), patients must have NSCLC with c-MET overexpression, MET amplification, or MET exon 14 skipping by local biomarker assessment as defined in study protocol. The number of patients with only c-MET overexpression is limited to 50% of enrolled patients in that dosing cohort including escalation and extension.
6. Progressive disease:

   a. Phase 1: Progressive disease on established standard medical anti-cancer therapy for his/her tumor type or intolerant to such therapy, or in the opinion of the investigator considered ineligible for a particular form of standard therapy on medical grounds.
7. At least one measurable lesion per response evaluation criteria in solid tumors (RECIST) 1.1, with the exception of bone-only disease (i.e., non-measurable disease per RECIST 1.1) with at least 1 radiological non-target lesion.
8. If not menopausal or surgically sterile, willing to practice at least one of the following highly effective methods of birth control for at least a (partner's) menstrual cycle before and for 3 months after study drug administration:

   1. True abstinence, when this is in line with the preferred and usual lifestyle of the patient, from sexual intercourse with a member of the opposite sex,
   2. Sexual intercourse with vasectomized male/sterilized female partner,
   3. Hormonal female contraceptive (oral, parenteral, intravaginal, implantable or transdermal) for at least 3 consecutive months prior to investigational product administration (when not clinically contraindicated as in breast, ovarian and endometrial cancers),
   4. Use of an intrauterine contraceptive device.
9. Resolution of prior-therapy-related AEs (including immune-related AEs but excluding alopecia) to ≤ Grade 1 per CTCAE, and no treatment for these AEs for at least 2 weeks prior to the time of enrollment. Alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 AEs not constituting a safety risk based on investigator's judgment are acceptable.
10. Phase 1 only: minimum of 2 weeks since last dose of hormone therapy.
11. Minimum of > 2 weeks or > 5 half-lives (whichever is longer) between the start of study treatment since last dose of radiotherapy, chemotherapy, or molecularly targeted agents or tyrosine kinase inhibitors; minimum of > 3 weeks of the start of study treatment since last dose of immunotherapy/monoclonal antibodies; > 6 weeks of the start of study treatment since the last dose of nitrosoureas, antibody-drug conjugates or radioactive isotopes.
12. Adequate organ function as indicated by the laboratory values.
13. Tissue and/or blood specimens:

    a. Phase 1: Available archival formalin-fixed, paraffin-embedded tumor tissue specimen.

    The archival tissue must be:
    * collected after progression from most recent prior systemic anti-cancer treatment, OR
    * the samples of previous lines of treatment. If patient wants to participate to the study but does not want to give the blood and tissue samples for the exploratory study, patient might be able to participate after discussion and approval of sponsor and the medical monitor.
14. If the patient agrees to optional pre- and/or study new tumor biopsies (that can be biopsied based on investigator's assessment) and to provide the tissue for biomarker analysis, a signed informed consent for the biopsy is required. Tissue obtained for the biopsy must not be previously irradiated. No systemic antineoplastic therapy may be received by the patient between the time of the biopsy and the first administration of ABN401.

    For escalation, each dose escalation cohort must try to enroll at least 1 patient who agrees to biopsies. An exception to the requirement for a new tumor biopsy in at least one patient per dose level is that if the first patient in a single dose cohort does not consent to a new tumor biopsy and the cohort is not expanded to 3 or 6 patients, a biopsy will not be required in that cohort. Note: During pre-treatment FFPE tissue samples (unstained slides or blocks) or new frozen tissue may be provided for tumor analyses.
15. Able and willing to comply with the protocol and the restrictions and assessments therein.

Exclusion Criteria:

1. Previous severe hypersensitivity reaction to any component of ABN401.
2. Prior therapy:

   a. Phase 1: Treatment with more than 4 lines of prior systemic therapy for recurrent/metastatic disease. If the patient was treated with more than 4 lines but his/her condition is eligible to participate to the trial by the investigator's judgement, the patient might be able to be enrolled to the trial under the medical monitor and the sponsor's approval,
3. Genetic analysis:

   a. Phase 1 Extension Cohort, existing data by genetic analysis of the patient's tumor tissue that may result in an increased probability of being resistant to c-MET inhibitors, including 1) EGFRi; 2) ALKi; 3) ROSi; 4) BRAFi; 5) NTRKi; 6) RETi,
4. Chronic inflammatory liver condition. History or clinical evidence of any liver or biliary pathology including cirrhosis, infectious disease, inflammatory conditions, steatosis, or cholangitis (including ascending cholangitis, primary sclerosing cholangitis, obstruction, perforation, fistula of biliary tract, spasm of sphincter of Oddi, biliary cyst or biliary atresia).
5. Prior organ or stem cell transplant.
6. Known active infection with HIV, HTLV-1, hepatitis B virus (HBV), or hepatitis C virus (HCV):

   1. Patients with a history of hepatitis B or C are allowed if HBV DNA or HCV RNA are undetectable,
   2. Active infection with human immunodeficiency virus (HIV) and CD4+ T-cell count <350/μL. Patients not on established ART for at least four weeks and having a detectable HIV viral load.
7. Symptomatic ascites or pleural effusion, unless clinically stable for at least two weeks following treatment for these conditions (including therapeutic thoraco- or paracentesis).
8. Known active CNS primary tumor or metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks prior to first dose of study drug, have no evidence of new or enlarging brain metastases and are off steroids for at least 15 days prior to first dose of study drug.
9. Known history of a hematologic malignancy, malignant primary brain tumor, or of a second malignant primary solid tumor (other than that under study), unless the patient has undergone potentially curative therapy with no evidence of that disease for 3 years. Note: The time requirement for no evidence of disease for 3 years does not apply to patients who underwent successful definitive resection of non-melanoma skin cancer, superficial bladder cancer, in situ cervical cancer, or other in situ cancers.
10. Active infection requiring therapy. However, subject with minor infections where oral antibiotic required, (e.g., urinary tract infection, Upper respiratory tract infection, etc.) could be eligible based on investigator's judgement.
11. Use of systemic corticosteroids > 10 mg/day prednisone or equivalent within 30 days or other immunosuppressive drugs within 30 days prior to first drug administration.
12. Received an investigational product or been treated with an investigational device within 30 days prior to first drug administration.
13. Has been receiving: radiotherapy, chemotherapy, or molecularly-targeted agents or tyrosine kinase inhibitors within 2 weeks or 5 half-lives (whichever is longer) of the start of study treatment; immunotherapy/monoclonal antibodies within 3 weeks of the start of study treatment; nitrosoureas, antibody-drug conjugates, or radioactive isotopes within 6 weeks of the start of study treatment; 7-day washout is permitted for palliative radiation (i.e. limited field, ≤ 14-day course of radiotherapy) to non-CNS lesions.
14. History or clinical evidence of any surgical or medical condition which the investigator judges as likely to interfere with the results of the study or pose an additional risk in participating e.g., rapidly progressive or uncontrolled disease involving a major organ system-vascular, cardiac, pulmonary, gastrointestinal, gynecologic, hematologic, neurologic, neoplastic, renal, endocrine, autoimmune or an immunodeficiency, or clinically significant active psychiatric or abuse disorders.
15. Is a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
16. Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study.
17. Patients with a corrected QT interval (using Fridericia's correction formula) (QTcF) of >470 msec (females) and >450 msec (males).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ABN401. | Measurements at Baseline till the last day of Visit
  Safety and tolerability determined by abnormal clinical laboratory tests, vitals signs, physical exam, ECG parameters, Liver function tests
To determine the objective response rate (ORR) to ABN401 according to RECIST 1.1 | Up to 30 days
  Objective response rate (ORR) is defined as the proportion of patients who experience a complete response (CR) or partial response (PR) as measured by RECIST 1.1.

SECONDARY OUTCOMES:
To determine the systemic PK of ABN401. | Dose Escalation Phase: Cycle 1- Day 1, Day 2, Day 5, Day 8, Day 15; Dose Expansion Phase: Cycle 1, Day -2, Day 1, Day 2, Day 8, Day 15
To determine preliminary estimate of ABN401 efficacy in patients with selected malignancies | Screening and at every 6 weeks from C1D1 independent of cycle length
  Efficacy will be assessed by CT/MRI Scans of the chest, abdomen and pelvis (patients with lung, pancreatic and ovarian cancer, and if clinically indicated for patients with other malignancies)
Evaluate the duration of response (DoR) to ABN401 according to RECIST 1.1 | Up to 30 days
  Duration of response (DoR) is defined as the time period from documentation of disease response to disease progression.
Assess the objective disease control rate (DCR) of ABN401 according to RECIST 1.1 | Up to 30 days
  Disease advanced control rate (DCR) is defined as the proportion of patients who achieve CR, PR, and stable disease (SD) as measured per RECIST 1.1.
Determine progression free survival (PFS) according to RECIST 1.1 | Up to 30 days
  Progression-free survival (PFS) is defined as the time from first dose of study drug until disease progression or death.

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (4):
  - ST George Private Hospital, Kogarah, New South Wales
  - Sydney Southwest Private Hospital, Liverpool, New South Wales
  - Scientia Clinical Research, Randwick, New South Wales
  - Linear Clinical Research, Perth, Western Australia
- South Korea (3):
  - National Cancer Centre, Goyang-si, Gyeonggi-do
  - Yonsei University Health System, Severance, Seoul
  - Asan Medical Centre, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://abionbio.com/